CLINICAL TRIAL: NCT04837794
Title: Self-Management of Chronic Pain Using a Digital Pain-Management Tool
Brief Title: Self-Management of Chronic Pain
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: University of California, San Diego (Other); PainDrainer AB (Industry)
Responsible Party: Sponsor
Other Study IDs: US1
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain
Keywords: self management; e-health; health tech; Digital Pain-Management Tool
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Digital Pain-Management Tool — Digital Pain-Management Tool

SUMMARY:
The investigators aim to validate if a digital tool for increased self-management of chronic pain can improve the quality of life for patients with chronic pain. The validation is based on the change in pain interference (Quality of life), pain intensity, physical functioning, depression, and anxiety based on self-reported information from baseline to study end.

DETAILED DESCRIPTION:
Chronic pain is today an increasing health problem in both Europe and US, with an estimation of about 90 million people affected in Europe (Breivik, H. et al., 2006) and 100 million people in US (Relieving Pain in America, IOM Report 2011), or 20-30% of the adult population around the world. Chronic pain is defined as a condition that lasts for at least three to six months, after the normal healing period of an injury. Medical interventions offered in clinics around the globe are unfortunately not giving the results needed to give back the quality of life the patients had prior to the onset of the pain. The treatments offered today do sometimes reduce pain, but the effect is minor, and new treatment regimens are needed (Relieving Pain in America, 2011). Recent quality assurance registry measurements in Sweden has shown that patient taken part of multi modal treatment regimens, such as the acceptance and commitment therapy, (ACT) show that less then 40% of the patients have a decline in the pain level of 1 level on the VAS scale, 55% has no effect and 9 % has an increased level of pain after going through the program (Nationel Register for Pain Rehabilitation, Sweden 2017) The study objective is to evaluate how the use of a digital pain coach, based on artificial intelligence that improves the self-management of pain will decrease the pain interference and thereby increase QoL among chronic pain patients, as measured by PROMIS pain interference 6a. We will here compare the improvement of quality of life by a decrease in pain interference, measured by PROMIS, in patients who follow their traditional treatment plan provided by the Pain Clinic with the addition of using a web application for increased self management of pain. The theory behind the study and the development of the device is supported by previously known data, showing that self-management has an effect and is important to the treatment by helping patients to believe in their own capacity to control their pain.

The present investigation aims at exploring the effect of including digital tool as an add on to standard treatment and rehabilitation and will measure the effect it has on:

Decreased pain interference Improved management of long-term pain and its consequences. Hence self-management of pain Increased function in daily life with the best possible activity and participation level Improved experience of health-related quality of life Decreased pain experience

ELIGIBILITY:
Inclusion Criteria:

* Have a complex, prolonged (neck shoulder pain or lower back pain
* Have been followed by a pain management specialist for at least 6 months
* Referred for Pain Medicine Consultation
* Be >18 years of age
* Be able to travel to and from the clinic
* Have a goal and motivation that is adequate in relation to the program offered
* Be medically prepared and not have any other medical examination or ongoing disease that constitutes an obstacle as well as adequate pharmacological treatment
* Have no major change in pain management (e.g. medications)
* Own a smart phone, tablet or computer or have the knowledge to use one

Exclusion Criteria:

* Low back pain requiring surgical intervention in the next 3 months
* Severe or acute psychiatric illness, severe anxiety or depression
* Reported/acute psychiatric illness or acute crisis
* Ongoing abuse of alcohol, drugs and drug-based drugs. This also includes high doses of prescribed drugs
* Pain related to malignancy
* Other areas of pain exceeding the level/intensity of low back or neck pain
* Currently involved in a lawsuit or pending litigation in relation to the low back or neck pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic pain patients at the UCSD Health System- Center for pain Medicine
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Pain interference | 6 and 12 weeks from baseline
  Change from baseline in pain interference (QoL), measured by PROMIS Pain Interference 6a . Measure of the amount of interference pain causes in life; range 6-30; higher is worse

SECONDARY OUTCOMES:
Pain severity | 6 and 12 weeks from baseline
  Change from Baseline in the 7 day average pain intensity. Measured by NRS using an 11-point Pain Intensity Numerical Rating Scale (NRS) (0=no pain, 10=pain as bad as you can imagine)
Physical function | 6 and 12 weeks from baseline
  Change from baseline in physical function, measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Physical function 10a.
  Measure of the impact of a condition on physical function; range 4-20; higher is worse
Depression | 6 and 12 weeks from baseline
  Change from Baseline measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression 4a.
  Measures the extent to which patients experience depressive symptoms over the past 7 days. Raw scores range from 4-20 with lower scores representing less endorsement of depression
Anxiety | 6 and 12 weeks from baseline
  Change from Baseline measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Anxiety 4.
  Measures the extent to which patients experience anxiety symptoms over the past 7 days. Raw scores range from 4-20 with lower scores representing less endorsement of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory R Polston, MD, Principal Investigator — UC San Diego Health
Locations (1):
- UC San Diego Health - Koman Family Outpatient Pavilion, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No